CLINICAL TRIAL: NCT00518375
Title: A Comparative, Open-label Study to Evaluate Graft Function in de Novo Renal Allograft Recipients Treated With Either a 'Reduced Dose' or a 'Standard Dose' of Cyclosporine in Combination With Sirolimus and Corticosteroids
Brief Title: Study Comparing Graft Function in Renal Allograft Recepients Receiving Reduced or Standard Dose CsA With Sirolimus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468E1-100154
Record Dates: First submitted 2007-07-27; First posted 2007-08-20 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2007-08

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Sirolimus; Cyclosporine; Adrenal Cortex Hormones

INTERVENTIONS:
Drug: Rapamune® (Sirolimus)
Drug: Neoral® (Cyclosporine)
Drug: Corticosteroids — Left up to local practice but steroids are typically used perioperatively

SUMMARY:
This study evaluated renal graft function (based on calcuated creatinine clearance) 12 months after transplantation in patients receiving either a regimen of reduced dose or standard dose cyclosporine in combination with sirolimus and corticosteroids. The incidence of acute graft rejection at 6 and 12 months following transplantation and patient and graft survival at 12 months were evaluated also.

DETAILED DESCRIPTION:
This study evaluated renal graft function (based on calcuated creatinine clearance) 12 months after kidney transplantation in patients receiving either a regimen of reduced dose or standard dose cyclosporine (CsA) in combination with sirolimus and corticosteroids. The incidence of acute graft rejection at 6 and 12 months following transplantation and patient and graft survival at 12 months after transplantation were evaluated also.

ELIGIBILITY:
Inclusion Criteria:

* Adults more than 18 years of age
* End-stage renal disease, with patients receiving a primary or secondary renal allograft from a cadaveric, living-unrelated or living-related mismatched donor
* Patients with a secondary transplant must have maintained their primary graft for at least 6 months

Exclusion Criteria:

* Planned antibody induction therapy
* Multiple organ transplants
* Patients at a high risk of acute rejection

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2000-04; Study Completion 2001-05

PRIMARY OUTCOMES:
Calculated creatinine clearance to evaluate renal function at 12 months post transplantation | 12 months

SECONDARY OUTCOMES:
Incidence of acute graft rejection at 6 and 12 months post transplantation and patient and graft survival at 12 months post transplantation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer